CLINICAL TRIAL: NCT06771999
Title: Attitudes Towards Deprescribing of Non-oncologic Medication in Cancer Pacient and the Impact of an Educational Intervention by a Clinical Pharmacist
Brief Title: Attitudes Towards Deprescribing Medications in Cancer Patients and Impact of Educational Intervention by a Clinical Pharmacist
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Mihaela Onea, PhD student, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 198/11OCT2024
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cancer Patients in Palliative Care with Chronic Use of Non-oncologic Medications
Keywords: palliative care; cancer; clinical pharmacist; educational intervention; rPATD
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: All participants will respond to two questionnaires, both validated in Romanian and some demographic information. One is the rPATD questionnaire that investigate attitudes towards deprescribing of medication and the other one is the HLS-EU-Q16 that investigates medical literacy of participants. After completion, the clinical pharmacist will give a brochure and a video about the process of deprescribing, information about the efficacy and the adverse reactions of medicines and the role of pacient in treatment decision. When participants come to another cancer treatment (after 14, 21 or 28 days), the rPATD will be completed again.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Educational intervention by a clinical pharmacist (Experimental): educational intervention using a brochure and a video with information about deprescribing, effectiveness and adverse reactions of medicines and the role of patient in treatment decision
  Interventions: Other: Educational intervention by a clinical pharmacist

INTERVENTIONS:
Other: Educational intervention by a clinical pharmacist — All participants will respond to two questionnaires, both validated in Romanian and some demographic information. One is the rPATD questionnaire that investigate attitudes towards deprescribing of medication and the other one is the HLS-EU-Q16 that investigates medical literacy of participants. After completion, the clinical pharmacist will give a brochure and a video about the process of deprescribing, information about the efficacy and the adverse reactions of medicines and the role of pacient in treatment decision. When participants come to another cancer treatment (after 14 , 21 or 28 days), the rPATD will be completed again.

SUMMARY:
Your participation in this study consists in responding to some questions from two questionnaires in Romanian about how you feel about deprescribing, your treatment and how you understand medical information. After that, you'll receive a brochure and watch a video with some basic information about medications and your involvement in treatment decisions and in the next visit for your cancer treatment you will be asked to answer questions from one of the initial questionnaire.

DETAILED DESCRIPTION:
Cancer patients are susceptible to using a lot of medications, with an increased risk of drug-related problems that could lead to adverse reactions from oncological drugs, hospital admissions, deteriorated performance status and increased mortality. In time, some medications may no longer be efficient, may have adverse reactions or may lose their indication and need to be stopped or replaced. This process is named deprescribing and it's supervised by a health care professional. Deprescribing can't be done without the implication of the patients, that's why it's important to investigate cancer patient's attitudes towards deprescribing non-oncologic medications in Romanian patients using a validated questionnaire (rPATD). Recent studies from Romania showed a possible lack of health care literacy that could affect patients involvement in treatment decision. In this study, we will investigate health care literacy using a validated questionnaire in Romanian (HLS-EU-Q16). In this study we will also investigate if an educational intervention (targeting patients involvement in treatment decision and mandatory, minimal information about efficacy of a treatment and its adverse reactions) conducted by a clinical pharmacist using a brochure and a video will improve their engagement and knowledge about drugs. Impact of educational intervention will be investigated by applying the rPATD questionnaire before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients in palliative treatment
* ECOG 1-2

Exclusion Criteria:

* cancer patients in curative treatment
* ECOG 3-4
* cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-13 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Impact of educational intervention performed by clinical pharmacist | from enrollment to the next cycle of oncological treatment (14, 21 or 28 days days)
  Participants will be asked to complete the same questionnaire before and after an educational intervention in order to assess if this kind of educational intervention is suitable for Romanian participants. Based on answers given to the same questions before and after the intervention, we can see if and what is changed in the perception of participants.

SECONDARY OUTCOMES:
Attitudes towards deprescribing medications in cancer patients in palliative treatment | from enrollment to the next cycle of oncological treatment (14, 21 or 28 days days) when they answer the second time
  Using the rPATD questionnaire (revised Patients Attitudes Towards Deprescribing ), we assess if Romanian cancer patients are willing to have their medication deprescribed
The level of health literacy | at enrollment
  Using the questionnaire HLS-EU-Q16 we can asses the level of health literacy of participants

OTHER OUTCOMES:
Demographic characteristics of the population included in this study | at enrollment
  We will be able to characterize a population of cancer patients in Romania (number of medications, number of diseases, social background, literacy)

CONTACTS AND LOCATIONS:
Locations (1):
- Constantin Opris Emergency County Hospital, Baia Mare, Maramureş, Romania

IPD SHARING:
Plan to Share IPD: Undecided
PhD contract might affect sharing the IPD until PhD defense

REFERENCES:
- [Background] Reeve E, Low LF, Shakib S, Hilmer SN. Development and Validation of the Revised Patients' Attitudes Towards Deprescribing (rPATD) Questionnaire: Versions for Older Adults and Caregivers. Drugs Aging. 2016 Dec;33(12):913-928. doi: 10.1007/s40266-016-0410-1. PMID 27785734
- [Background] Linsky A, Gellad WF, Linder JA, Friedberg MW. Advancing the Science of Deprescribing: A Novel Comprehensive Conceptual Framework. J Am Geriatr Soc. 2019 Oct;67(10):2018-2022. doi: 10.1111/jgs.16136. Epub 2019 Aug 20. PMID 31430394
- [Background] Coman MA, Forray AI, Van den Broucke S, Chereches RM. Measuring Health Literacy in Romania: Validation of the HLS-EU-Q16 Survey Questionnaire. Int J Public Health. 2022 Feb 4;67:1604272. doi: 10.3389/ijph.2022.1604272. eCollection 2022. PMID 35185446
- [Background] Bucsa C, Onea M, Rusu A, Farcas A, Porojan M, Dumitrascu D, Iaru I, Leucuta D, Mogosan C, Reeve E, Moga D. Translation, cultural adaptation and validation of the revised patients' attitudes towards deprescribing (rPATD) questionnaire in Romanian older adults. Res Social Adm Pharm. 2023 Nov;19(11):1471-1479. doi: 10.1016/j.sapharm.2023.07.011. Epub 2023 Jul 20. PMID 37495451
- [Background] Whitman A, DeGregory K, Morris A, Mohile S, Ramsdale E. Pharmacist-led medication assessment and deprescribing intervention for older adults with cancer and polypharmacy: a pilot study. Support Care Cancer. 2018 Dec;26(12):4105-4113. doi: 10.1007/s00520-018-4281-3. Epub 2018 Jun 4. PMID 29869294